CLINICAL TRIAL: NCT06682299
Title: Transitioning From Maintenance ECT to Maintenance TMS in Treatment Resistant Depression
Brief Title: Maintenance TMS in Treatment Resistant Depression
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Austin Messner (Other)
Responsible Party: Sponsor-Investigator, Austin Messner, Senior Medical Resident, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 95789
Record Dates: First submitted 2024-11-07; First posted 2024-11-12 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-04

CONDITIONS: Treatment Resistant Depression (TRD)
Keywords: depression; tms; ect; treatment resistant depression; trd
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant; Depression; Epilepsy, Rolandic

STUDY DESIGN:
Intervention Model Description: Open label patient preference trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- TMS (Experimental): Patients who have achieved remission of treatment resistant depression through an initial course of ECT (8 to 12 sessions) at the University of Kentucky will be identified by the ECT attending physician as a candidate for this study. They will receive TMS in this arm of study for maintenance treatment of their depression and monitored with depressive scales.
  Interventions: Device: Transmagnetic Stimulation
- ECT (Active Comparator): Patients who have achieved remission of treatment resistant depression through an initial course of ECT (8 to 12 sessions) at the University of Kentucky will be identified by the ECT attending physician as a candidate for this study. If they elect to continue with maintenance ECT treatments which is the current standard of care, their depressive symptoms and cognitive functioning will be monitored accordingly.
  Interventions: Device: Electroconvulsive Therapy

INTERVENTIONS:
Device: Transmagnetic Stimulation — TMS will be given for the maintenance treatment of treatment resistant depression following successful course of ECT (8-12 treatments).
  Other Names: TMS
  Arms: TMS
Device: Electroconvulsive Therapy — Patients will remain in standard of care treatment and receive maintenance ECT treatments for treatment resistant depression
  Other Names: ECT
  Arms: ECT

SUMMARY:
Electroconvulsive therapy (ECT) is one of the most efficacious treatments available for treatment-resistant depression (TRD). Although a maintenance ECT protocol exists, multiple barriers limit its use for long-term use. These barriers include procedure tolerability, cognitive side effects, financial burden, and unreliable social support to accompany patients for these treatments. On the other hand, a different modality of noninvasive neuromodulation called transcranial magnetic stimulation (TMS) can be performed in the outpatient setting and does not need anesthesia. The likelihood of cognitive adverse effects with TMS is much lower than with ECT. Our clinical question encompasses piloting a maintenance TMS regimen to maintain remission in treatment-resistant major depressive disorder.

This will be a patient-preference clinical trial, with patients offered the choice to initiate maintenance TMS versus maintenance ECT after their index ECT sessions for treatment-resistant depression. There will be no randomization or placebo involved in this study.

DETAILED DESCRIPTION:
The clinical question encompasses piloting a maintenance TMS regimen to maintain remission in treatment-resistant major depressive disorder.

Patients who choose maintenance TMS will initiate maintenance TMS sessions on day one of the study and continue any currently prescribed pharmacotherapy. Participants will initiate TMS treatment within 1 week of last index ECT treatment. Participants will then follow a schedule of weekly for 4 sessions, every other week for 4 sessions, and monthly for 3 sessions for a total of 11 sessions in 6 months. Investigators will use the TMS paradigm called intermittent theta burst stimulation (iTBS), which was used in the SNT trial(Cole et al., 2022; Cole et al., 2020). At conclusion of the 6 month TMS portion of the study clinical judgement will be used to determine if the patient will return to maintenance ECT treatment. RBANS for assessment of cognition will be completed at the beginning, after 6 months, and at the conclusion of the study as well in both the standard of care and TMS portions of the study.

Those who choose maintenance ECT will transition to maintenance ECT treatments in the hospital as prescribed by their treating inpatient psychiatrists. On initial visit consent will be obtained and baseline cognitive and behavioral scales assessed as follows: Antidepressant treatment history form (ATHF), alcohol use disorder identification test (AUDIT-C), Hamilton Depression Rating Scale (HDRS), Clinical Global Impression (CGI), quick inventory of depressive symptomology (QIDS), Brief Psychiatric Rating Scale (BPRS), Drug Abuse Screening Test (DAST-10), Repeatable Battery for the Assessment of Neuropsychological Status Update (RBANS), standardized assessment of personality abbreviated scale (SAPAS). Patients will then be asked to return at 6 month and 12 month intervals to repeat HDRS, QIDS, RBANS, and CGI scales.

Research data will be collected primarily through self assessment scales including Antidepressant treatment history form (ATHF), alcohol use disorder identification test (AUDIT-C), Hamilton Depression Rating Scale (HDRS), Clinical Global Impression (CGI), quick inventory of depressive symptomology (QIDS), Brief Psychiatric Rating Scale (BPRS), Drug Abuse Screening Test (DAST-10), Repeatable Battery for the Assessment of Neuropsychological Status Update (RBANS), standardized assessment of personality abbreviated scale (SAPAS).

ELIGIBILITY:
Inclusion Criteria:

* Patients treated for TRD who have achieved remission through an index series of ECT
* Able to provide informed consent
* Age between 18 and 65 years
* Deemed appropriate for maintenance TMS by their psychiatrist
* Right-handed

Exclusion Criteria:

* History of seizures or a seizure disorder
* Related neurological disorder, or any other medical condition that would preclude TMS treatment determined by the treatment team.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-04-17 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Change in Hamilton Depression Rating Scale (HDRS) | Baseline and prior to each procedure for duration of study, up to six months
  One of the most widely used clinician administered depression scales containing 17 items. Scores range from 0 to 54 with 0-7 being normal, 8-16 being mild depression, 17-23 moderate depression and 24 or greater being severe depression. Higher scores equate to more severe depressive symptoms.

SECONDARY OUTCOMES:
Change in Quick inventory of depressive symptomatology (QIDS) | Baseline and prior to each procedure for duration of study, up to six months
  A widely used self-report scale of depression with similar validity to the HDRS that consists of 16 scale items. Scores range from 0 to 27 with 0-5 indicating no depression, 6-10 mild depression, 11-15 moderate depression, 16-20 severe, and 21 or higher very severe. Higher scores equate to more severe depressive symptoms.
Change in Repeatable Battery for the Assessment of Neuropsychological Status Update (RBANS) | Baseline on initial presentation, at 6 months, and at 12 months
  Cognitive screening tool that is individually administered battery to measure cognitive decline or improvement. Scores range from 40 to 160. 69 and below is extremely low, 70-79 borderline, 80-89 low average, 90-109 average, 110-119 high average, 12-129 superior, and 130+ very superior. Higher scores equate to better cognitive functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Gopalkumar Rakesh, MD, Study Director — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Rachid F. Safety and Efficacy of Theta-Burst Stimulation in the Treatment of Psychiatric Disorders: A Review of the Literature. J Nerv Ment Dis. 2017 Nov;205(11):823-839. doi: 10.1097/NMD.0000000000000742. PMID 29077650
- [Background] Rossi S, Hallett M, Rossini PM, Pascual-Leone A; Safety of TMS Consensus Group. Safety, ethical considerations, and application guidelines for the use of transcranial magnetic stimulation in clinical practice and research. Clin Neurophysiol. 2009 Dec;120(12):2008-2039. doi: 10.1016/j.clinph.2009.08.016. Epub 2009 Oct 14. PMID 19833552
- [Background] Wilson S, Croarkin PE, Aaronson ST, Carpenter LL, Cochran M, Stultz DJ, Kozel FA. Systematic review of preservation TMS that includes continuation, maintenance, relapse-prevention, and rescue TMS. J Affect Disord. 2022 Jan 1;296:79-88. doi: 10.1016/j.jad.2021.09.040. Epub 2021 Sep 17. PMID 34592659
- [Background] Magnezi R, Aminov E, Shmuel D, Dreifuss M, Dannon P. Comparison between neurostimulation techniques repetitive transcranial magnetic stimulation vs electroconvulsive therapy for the treatment of resistant depression: patient preference and cost-effectiveness. Patient Prefer Adherence. 2016 Aug 4;10:1481-7. doi: 10.2147/PPA.S105654. eCollection 2016. PMID 27536079